CLINICAL TRIAL: NCT01511354
Title: Development of New Stable Isotope Method to Determine Protein Requirements in Critically Ill Children
Brief Title: New Stable Isotope Method to Determine Protein Requirements in Critically Ill Children
Status: Completed | Type: Observational
Sponsor: Texas A&M University (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Other Study IDs: 101653
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Critically Ill
Keywords: critically ill children; ICU; 24hr protein balance; stable isotopes; fed state
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard clinical care: Standard nutritional therapy and treatment

SUMMARY:
The need for certain components of food (i.e. protein) for critically ill children is not clear. It is important to have critically ill children fed adequately to prevent that their condition becomes worse or that recovery takes longer. Research methods used in the past to investigate the need for protein (Nitrogen Balance calculations), were not sensitive enough in severely ill children. The purpose of this study is to develop a new research method to determine the need for protein in severely ill children. In order to develop this new method, more information is needed on the way the body of these children uses protein in 24-hours. In the present study during 24-hours 8 children of age less than 18 years who are admitted to either the Pediatric ICU or the Cardiovascular ICU. Subjects will receive a standard nutrition, providing an age specific amount of protein (age ≤ 3: 2.52 protein g/kg BW.d; age 4-6: 1.8 protein g/kg BW.d; age > 10: 1.44 protein g/kg BW.d) via tube feeding. They will also receive a mixture of stable isotopes of amino to investigate protein behavior in the body (protein kinetics) both by infusion in their blood and together with the nutrition. Blood will be drawn every 60 minutes during the 24-hour period and the behavior of protein and the concentrations in blood of amino acids and urea will be measured. Urine will be collected to measure nitrogen balance. The investigators will compare the results of this nitrogen balance method with the results of the stable isotope method. PIM2, PRISM, SIRS criteria will be used to get information on the severity of illness of the subjects. Also body weight and length as well as body composition of the subjects will be measured at the start and after the 24-hour period. Body composition will be measured by Bioelectrical Impedance Spectroscopy. Endpoints of the study are net whole-body protein synthesis (protein balance), 24-hour pattern of protein balance, 24-hour urea production, 24-hour nitrogen balance, 24-hour contribution of arginine kinetics to whole body protein breakdown, 24-hour muscle protein breakdown, splanchnic amino acid extraction and plasma amino acid concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill children with age less than 18 years at the time of enrollment
2. Admitted to the Pediatric ICU or Cardiovascular ICU, with an expected stay of >72 hours
3. One arterial line (or umbilical arterial line) and one multi-lumen central venous line (or two peripheral venous catheters) in place.
4. Continuous total parenteral nutrition or continuous enteral feeding (e.g. via nasogastric, nasoduodenal, gastric, jejunal tube) with standard nutrition appropriate for age and weight expected during admission.
5. No planned major changes or interventions (such as surgery) in the treatment and care of the patient from enrollment to completion of study period (end of 24-hour stable isotope infusion protocol).
6. Hemodynamic stable condition (with or without continuous inotropic medication) defined as ≤1 boluses of volume resuscitation for hypotension in 24 hour.
7. No significant loss of plasma/blood from wounds or drains, that may influence the results of the study, no chylothorax.
8. Informed consent by parent(s) or LAR.

Exclusion Criteria:

1. Congenital/acquired metabolic or endocrine disorders or hepatic or renal failure or anuria or oliguria.
2. Gastrointestinal obstructions or any condition that causes malabsorption.
3. Active gastro-intestinal bleeding.
4. Fluid restriction (<100 ml/kg BW.day) making administration of intravenous and enteral stable isotopes impossible.
5. Any other condition that according to the Principal Investigator or study physician would interfere with collecting study samples (for example isolation due to MRSA infection).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Stable critically ill children admitted to the Pediatric Intensive Care Unit or Cardiovascular Intensive Care Unit of ACH
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Whole body protein synthesis rate | 24 hours
  Whole body protein synthesis rate in the fed state

SECONDARY OUTCOMES:
Whole body protein breakdown rate | 24 hours
  Whole body protein breakdown rate in the fed state
Whole body protein breakdown rate | 24 hours
  Whole body myofibrillar protein breakdown rate in the fed state
Whole body Arginine production rate | 24 h
  Net whole body arginine production rate in the fed state
Splanchnic amino acid extraction | 24 hr
  Splanchnic amino acid extraction in the fed state
Urea production | 24 hr
  Whole body urea production in the fed state
Plasma amino acid levels | 24 hr
  Plasme amino acid level in the fed state

CONTACTS AND LOCATIONS:
Overall Officials: Marielle P Engelen, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] de Betue CTI, Garcia Casal XC, van Waardenburg DA, Schexnayder SM, Joosten KFM, Deutz NEP, Engelen MPKJ. 24-Hour protein, arginine and citrulline metabolism in fed critically ill children - A stable isotope tracer study. Clin Nutr. 2017 Jun;36(3):876-887. doi: 10.1016/j.clnu.2016.12.023. Epub 2017 Jan 4. PMID 28089618